#### MEDICAL RECORD

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

Adult Patient or

• Parent, for Minor Patient

INSTITUTE: National Cancer Institute

STUDY NUMBER: 18-C-0057 PRINCIPAL INVESTIGATOR: Raffit Hassan, M.D.

STUDY TITLE: A Phase I Study of the Mesothelin-Targeted Immunotoxin LMB-100 in Combination with

SEL-110 in Subjects with Malignant Pleural or Peritoneal Mesothelioma

Continuing Review Approved by the IRB on 01/07/19

Amendment Review Approved by the IRB on 10/04/18 (D)

Date posted to web: 01/17/19

Standard

#### INTRODUCTION

We invite you to take part in a research study at the National Institutes of Health (NIH).

First, we want you to know that:

Taking part in NIH research is entirely voluntary.

You may choose not to take part, or you may withdraw from the study at any time. In either case, you will not lose any benefits to which you are otherwise entitled. However, to receive care at the NIH, you must be taking part in a study or be under evaluation for study participation.

You may receive no benefit from taking part. The research may give us knowledge that may help people in the future.

Second, some people have personal, religious or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). If you have such beliefs, please discuss them with your NIH doctors or research team before you agree to the study.

Now we will describe this research study. Before you decide to take part, please take as much time as you need to ask any questions and discuss this study with anyone at NIH, or with family, friends or your personal physician or other health professional.

## Why is this study being done?

In this study, we will determine a safe dose of LMB-100 plus SEL-110 in patients with advanced mesothelioma. LMB-100 and SEL-110 are both investigational agents, meaning that they have not been approved by the US Food and Drug Administration. LMB-100 is a type of manufactured protein which is similar to protein normally produced by your body in response to a specific foreign substance. LMB-100 is attracted to the mesothelin protein, which is present in a lot of different tumors, including mesothelioma, but is found in only a very small number of

PATIENT IDENTIFICATION

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or

• Parent, for Minor Patient

NIH-2514-1 (07-09) P.A.: 09-25-0099

| MEDICAL RECORD | NIE | NTINUATION SHEET for either: I 2514-1, Consent to Participate in A Clinical Research Study I 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|---|
| STUDY NUMBER: | 18-C-0057 | CONTINUATION: pages |

normal tissues. After binding to the mesothelin on tumors, LMB-100 can then attack and kill cancer cells. However, sometimes the body creates substances (called antidrug antibodies – ADAs) that will attack LMB-100, which reduces how well it can work. It is thought that adding SEL-110, which is a nanoparticle that contains rapamycin (a drug used to prevent the rejection of transplants) will prevent the formation of ADAs.

## Why are you being asked to take part in this study?

You are being asked to take part in this study because you have pleural or peritoneal mesothelioma that has not responded to prior platinum based therapy.

## How many people will take part in this study?

Up to 23 patients will be enrolled on the study.

## **Description of Research Study**

You will receive LMB-100 through an IV catheter (a tube inserted in a vein, usually in your arm) on day 1, day 3 and day 5 of each 21-day cycle. SEL-110 will be given on day 1 of each 21-day cycle. You will receive LMB-100+SEL-110 for up to 4 cycles or until your disease worsens or you have intolerable side effects, whichever happens first. In the first part of the study (12 – 15 patients) we will test various dose combinations of LMB-100 and SEL-110. Depending on whether intolerable side effects occur in any group of 3-6 patients enrolled, we will adjust the doses of the drugs, testing each combination in 3 – 6 subjects until we find the maximum dose combination that does not cause intolerable side effects in too many subjects. Once a safe dose has been determined, an additional 6 patients will be enrolled at that dose. The dose you receive depends on when you enroll in the study.

Once you have finished taking the drugs, we would also like to follow you after you have finished taking the study drug to keep track of your disease status (progression) if this was not the reason you were removed from the study.

## Before you begin the study

Before beginning the study, you will need to have tests and/or procedures to help your doctor verify whether you can participate. This is called screening. Most of the exams, tests, and procedures you will have are part of the usual approach for your cancer. However, there are some extra procedures that you will need to have if you take part in this study. If you have already undergone some of these examinations very recently, your doctor may decide not to repeat them. Briefly, these tests, which are performed under a separate consent, include:

• Confirmation of diagnosis (You must provide a sample tumor tissue for an evaluation by the NCI Laboratory of Pathology. The tissue may be from a previous surgery, biopsy or collection from a tumor effusion (fluid around the tumor). If none is available, we will

PATIENT IDENTIFICATION CONTINUATION SHEET for either:

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 18-C-0057 CONTINUATION:  pages

ask you to have a biopsy or a collection of effusion material to provide a fresh sample). Please see page 9, Tumor Biopsies and Effusions for a description of the procedure.

- Medical history and physical examination
- Routine blood and urine tests including pregnancy test in women who can have children. Pregnant women will not be allowed on study.
- Scans and x-rays
- Electrocardiogram (ECG)
- Echocardiogram
- Tests for viruses (hepatitis and HIV)

## **During the study**

Once it is determined that you are eligible and you have signed the consent for the study, you will receive IV infusions of LMB-100 and SEL-110 as described above. Each SEL-110 infusion lasts about an hour and each LMB-100 infusion will last about 30 minutes, but it might take longer if your study doctor decides it is needed for your safety. On day 1 of each cycle, when both medications are given, you will receive the LMB-100 immediately after you have completed the SEL-110 infusion. You will be monitored for side effects for 2 hours after your first infusion of LMB-100, and for 30 minutes after all other infusions if no side effects occurred previously. We will give you standard pre-medications that include an antihistamine (such a Benadryl), acetaminophen (Tylenol), ranitidine (Zantac) and dexamethasone, a steroid to help prevent infusion related side effects.

While you are taking study medication, we will perform several tests and examinations for safety and to test the effect of the study therapy.

These include routine blood and urine tests that will be done 4-8 times per cycle, pregnancy tests for women that can have children once during each cycle, scans that will be performed approximately every 6 weeks, and ECGs that will be done before each LMB-100 infusion. Some of the laboratory tests may be done by your local lab or physician. Your study team will discuss which ones.

We will also perform tests for research studies to find out how your body handles the drugs (PKs), the types of immune cells present in your disease, how your body reacts to the drug and how certain side effects of the LMB-100 might be caused. Most of the sampling for these research tests will be done before your first dose of study drug, on the days you take the study drug (just before or just after you get the study drug) or at the end of treatment. In addition, a blood sample will be collected at the end of cycle 2 and on day 8 ( $\pm$  2 days) of each cycle. Exceptions to this are:

• PK studies on days 1 and 5 of cycle 1 and on day 1 of cycles 2 -4. These samples will be drawn before your infusion and periodically for up to 25 hours after the start of SEL-100

**CONTINUATION SHEET for either:** 

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | NII | NTINUATION SHEET for either: I 2514-1, Consent to Participate in A Clinical Research Study I 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|---|
| STUDY NUMBER: | 18-C-0057 | CONTINUATION: pages |

infusion on days 1 of cycles 1- 4 and 24 hours after the start of LMB-100 infusion on day

• Optional biopsies which may be collected before the first dose of LMB-100 (if you have not given a biopsy at screening) and after you have completed two cycles of therapy. The biopsies to be performed are exclusively for research purposes and will not benefit you. It might help other people in the future. You will be given the opportunity to decide whether you want to have these sample collected at the time of each biopsy. All tissue will be reviewed by the NCI Laboratory of Pathology.

*To be avoided during the study* 

1 of cycle 5.

- There are certain medications and foods known to interact with rapamycin that should be avoided from 14 days prior to your first dose of study therapy to the last dose SEL-110. These include grapefruit juice, St. John's wort, certain anti-fungal medications and calcium channel blockers. Please let your doctor know the medications that you are taking.
- Because rapamycin can reduce your white blood cells, you should avoid anyone that has an active infection

## When you are finished taking the drugs

You will be asked to return to the NIH for an end of treatment visit on the last day of cycle 4 and for a follow up visit approximately 6 – weeks after you have had your last dose of study drug to have the following tests:

- Medical history and physical exam
- Routine blood tests
- Pregnancy test if you are a woman who can have children (follow up visit only)
- Scans if your disease has not worsened since the beginning of the study
- ECG

If after this visit, your disease has not gotten worse, we would like to continue to scan you and perform blood tests every 6 weeks until your disease worsens; however, this is not required.

## **Birth Control / Pregnancy / Fertility**

If you are a woman who is breast feeding or pregnant, you may not take part in the study because we don't know how this medicine would affect your baby or your unborn child. Animal studies performed with an oral form of the active ingredient (a drug called rapamycin) contained in SEL-110 showed adverse effects when given to pregnant rats. These effects included death of the fetus, reduced fetal weights, and delays in the formation of bones. It is not known whether these effects would also occur in humans; however, a similar risk in humans should be considered

## PATIENT IDENTIFICATION CONTINUATION SHEET for either:

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | NI | ONTINUATION SHEET for either:<br>H 2514-1, Consent to Participate in A Clinical Research Study<br>H 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|---|
| STUDY NUMBER: | 18-C-0057 | CONTINUATION: pages |

possible. If you are a woman who can become pregnant, or are the partner of a woman who can become pregnant, you will need to practice an effective form of birth control before starting study treatment, during study treatment, and for three months after you finish study treatment. Men who are considering participation in this study should be aware that their ability to father a child might be impaired. Studies with SEL-110 administered to rats in three monthly doses by intravenous injection showed a decrease in the size of the testes and prostate in male rats, as well as a decrease in sperm count. It is not known whether the reduction of sperm count is reversible in rats. Among male patients taking an oral form of the active ingredient contained in SEL-110 (a drug called "rapamycin") that was given daily or three times weekly for the prevention of transplant rejection, those reporting low or no sperm counts after treatment for more than 6 months eventually achieved partial to full reversibility of sperm production after treatment ended. We do not know whether changes in sperm count would be reversed at similar rates after SEL-110 treatment is ended.

In addition, male subjects should not donate sperm during the study and for 3 months after the last dose of study therapy. If you think that you or your partner is pregnant, you should tell your study doctor or nurse at once.

Effective forms of birth control include:

- abstinence
- intrauterine device (IUD)
- hormonal [birth control pills, injections, or implants]
- tubal ligation
- vasectomy

## **Risks or Discomforts of Participation**

#### Risks and Possible Undesirable Effects of LMB-100

Prior to this study LMB-100 has only been given to 15 subjects; therefore, we do not know all of the possible side effects. However, below is a list of the most common and most serious side effects occurring on the earlier study, some occurring at higher doses than will be used in this study.

*The most common side effects (some were serious) were:* 

- Low levels of the blood protein albumin which may lead to swelling, muscle weakness or loss of appetite
- Tiredness
- Swelling of the arms and legs

#### **CONTINUATION SHEET for either:**

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

MEDICAL RECORD

CONTINUATION SHEET for either:

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 18-C-0057 CONTINUATION:  pages

- Nausea
- Fever
- Decreased appetite
- Shortness of breath
- Pain in muscles

Less common, but serious side effects included:

- Fluid in the organs which may cause low blood pressure, shortness of breath, swelling of ankles
- Abnormal heartbeat
- Reactions during or following the infusion of the drug which may cause fever, chills, rash or low blood pressure
- Pain in joints
- Kidney damage which may cause swelling, may require dialysis

## Other possible side effects

Other possible side effects discussed below are based on side effects that occurred when testing a similar agent, SS1P and in animal studies of LMB-100. It is possible that there may be other unexpected side-effects that occur in addition to those listed below.

LMB-100 may cause inflammation to membranes causing chest pain, shortness of breath, low blood pressure, and heart failure. In animals, some mild kidney toxicity was seen, characterized by increased enzymes and protein in the urine. This will be checked for with regular blood and urine tests.

As with other drugs similar to LMB-100, there is a chance that the drug could cause the body to produce an unwanted response called 'Anti-drug antibodies' (ADAs). These might not cause problems however there is a chance they could lead to a severe anti-drug response in the body. ADA levels will be measured during the study to monitor any changes.

There may also be pain and swelling at the infusion site.

It is important that you contact your doctor as soon as you experience any side effects whether you think the treatment has caused them or not. You must also tell your doctor if you have started any new medication or had a change to your existing medication. This includes medications available without a prescription (over the counter) and alternative medicines. If you have any questions or concerns about any of the information provided above, about the possible side effects of treatment, or the possible consequences of treatment for those side effects, please ask the principal investigator or the research staff for more information.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

MEDICAL RECORD

CONTINUATION SHEET for either:

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 18-C-0057 CONTINUATION:  pages

## The most important symptoms you need to report to your doctor <u>immediately</u> are:

- o possible infusion or allergic reactions (symptoms that start during or within a few hours of the infusion, e.g., wheezing, tightness in the throat or chest, rash, and facial swelling)
- o chest pain
- o shortness of breath
- o palpitations (fast heart beat)
- o bleeding and high fever
- o impaired brain function (e.g., dizziness, blurred vision, confusion)

If you experience any severe or dangerous side effect, you should:

- 1. Seek professional medical help immediately.
- 2. Call your study doctor.
- 3. If necessary, go to the nearest emergency room.

#### Risks and Possible Undesirable Side Effects of SEL-110

Potential risks included are those that have been identified in studies prior to being tested in humans, and from how well similar marketed (available) medications have been tolerated.

- <u>Infusion reactions</u>. Symptoms of infusion reaction may include the following: headache, nausea, dizziness, rash, body aches, fever, chills, fatigue, change in blood pressure, flushing (turning red) or tickling in your throat.
- Anaphylaxis is a potentially life threatening allergic reaction. Symptoms which may
  include the following: a change in blood pressure, coughing, wheezing, shortness of
  breath, itching around the mouth and/or tongue, swelling of lips and/or tongue, dizziness,
  passing out, skin hives, redness of skin, swelling of skin, vomiting, nausea, diarrhea, or
  cramps.
- <u>Damage to the lungs</u> which may cause shortness of breath a condition called pneumonitis
- Reduction in number of white blood cells a condition called Leukopenia.
- Opportunistic Infection if your immune system is weak, an infection may occur caused by bacteria, a virus, or a fungus, or parasites.
- <u>Disturbances to your metabolic system including:</u>
  - o Hyperglycemia- increase in blood sugar in the blood stream
  - o Hypertriglyceridemia- increase in triglycerides
  - o Hypercholesterolemia- increase in cholesterol
  - o Hypophosphatemia- low levels of phosphate in the blood

PATIENT IDENTIFICATION

#### **CONTINUATION SHEET for either:**

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 18-C-0057 CONTINUATION:  pages

- Gout Flares a worsening of your gout symptoms.
- <u>Methemoglobinemia</u> a blood disorder where abnormal amounts of methemoglobin, which is a form of hemoglobin, is produced.
- <u>Antibody Development</u> you may develop antibodies to the medication, which may decrease its effectiveness; or increase the likelihood of an allergic reaction.
- <u>Stomatitis</u> painful swelling and sores inside the mouth which may require medication to help them resolve.

You may or may not develop any of these symptoms during this study. There may be other risks that are unknown.

## **Risks from pre-medications**

## Acetaminophen

Acetaminophen is considered to be safe and effective in the recommended doses. However, when taken incorrectly acetaminophen can cause liver damage. Your risk of liver damage may be increased if you drink more than three alcoholic drinks every day, take more than the recommended dose (overdose), or if you take any additional drugs that also contain acetaminophen at the same time.

## Diphenhydramine

Drowsiness, dizziness, constipation, stomach upset, blurred vision, or dry mouth/nose/throat may occur when taking diphenhydramine.

#### Ranitidine:

It can cause constipation, diarrhea, headache, nausea or upset stomach. Rare serious side effects include severe allergic reaction with rash, hives, itching, difficulty breathing; confusion, dark urine, depression, fast or slow heartbeat, unusual bruising or bleeding, yellowing of the eyes or skin (indicating liver damage).

#### Dexamethasone:

Stomach upset, headache, dizziness, changes in your period, trouble sleeping, increased appetite, or weight gain may occur. Rarely patients using dexamethasone have experienced increased infection, bone/joint pain, thirst, increased urination, irregular heartbeat, eye pain, vision problems, black stools, vomit that looks like coffee grounds, puffy face, swelling of the feet and ankles, pain/redness/swelling of the arms or legs, tiredness, mood changes, unusual hair/skin growth, muscle cramps, weakness, easy bruising/bleeding, slow wound healing, thinning skin and seizures.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 18-C-0057 CONTINUATION:  pages

## **Risks from Study Procedures**

The following study procedures and treatments may have risks and cause discomfort while you participate on this study:

#### Blood draws

There is the risk of slight pain, bruising or infection when your blood is drawn. Drawing blood may cause some people to faint.

#### **ECGs**

The glue used to keep the electrodes in place during the ECG may irritate your skin and cause redness.

## Tumor Biopsies and Effusions

Tumor biopsies and tumor effusions: local anesthesia of the skin will be given prior to any tumor biopsy or effusion collection, in order to prevent painful sensations. However, you may still experience pain or discomfort at the biopsy site. Irritation, redness, swelling and/or bleeding may also occur. There is a risk of abnormal healing, fever, infection or of an allergic reaction to the anesthetic agent used to anesthetize the skin at the biopsy site. Once the sample has been obtained, a stitch may be used to close the wound and facilitate healing.

In some cases, we may use CT scans to help guide us during your biopsy. This introduces the added risk of research radiation. This research study may involve exposure to radiation from up to 2 CT guided tumor biopsies. This radiation exposure is not required for your medical care and is for research purposes only. The amount of radiation you will receive in this study is 1.6 rem which is below the guideline of 5 rem per year allowed for research subjects by the NIH Radiation Safety Committee. The average person in the United States receives a radiation exposure of 0.3 rem per year from natural sources, such as the sun, outer space, and the earth's air and soil. If you would like more information about radiation, please ask the investigator for a copy of the pamphlet, An Introduction to Radiation for NIH Research Subjects.

While there is no direct evidence that the amount of exposure received from participating in this study is harmful, there is indirect evidence it may not be completely safe. There may be a very slight increase in the risk of cancer.

Please tell your doctor if you have had any radiation exposure in the past year, either from other research studies or from medical tests or care, so we can make sure that you will not receive too much radiation. Radiation exposure includes x-rays taken in radiology departments, cardiac catheterization, and fluoroscopy as well as nuclear medicine scans in which radioactive materials were injected into your body.

| MEDICAL RECORD | CONTINUATION SHEET for either: NIH 2514-1, Consent to Participate in A Clinical Research Study NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|
|---|---|

STUDY NUMBER: 18-C-0057 CONTINUATION:  pages

## **Potential Benefits of Participation**

The aim of this study is to find a safe dose for this experimental treatment. We do not know if you will receive personal, medical benefit from taking part in this study. These potential benefits could include shrinking of your tumor or lessening of your symptoms, such as pain, that are caused by the cancer. Because there is not much information about the drug's effect on your cancer, we do not know if you will benefit from taking part in this study, although the knowledge gained from this study may help others in the future who have cancer.

## **Alternative Approaches or Treatments**

Instead of being in this study, you have these options:

- Getting treatment or care for your cancer without being in a study
- Taking part in another study
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly. Instead, it tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

Please talk to your doctor about these and other options.

## **Research Subject's Rights**

#### What are the costs of taking part in this study?

If you choose to take part in the study, the following will apply, in keeping with the NIH policy:

- You will receive study treatment at no charge to you. This may include surgery, medicines, laboratory testing, x-rays or scans done at the Clinical Center, National Institutes of Health (NIH), or arranged for you by the research team to be done outside the Clinical Center, NIH if the study related treatment is not available at the NIH.
- There are limited funds available to cover the cost of some tests and procedures performed outside the Clinical Center, NIH. You may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the Clinical Center, NIH.
- Once you have completed taking part in the study, medical care will no longer be provided by the Clinical Center, NIH.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | NIE | NTINUATION SHEET for either: I 2514-1, Consent to Participate in A Clinical Research Study I 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|---|
| STUDY NUMBER: | 18-C-0057 | CONTINUATION: pages |

Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The National Cancer Institute (NCI) and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Cancer Institute Institutional Review Board
- Qualified representatives from Selecta Biosciences, Inc., the pharmaceutical company who produces SEL-110.

A description of this clinical trial will be available on <a href="http://www.Clinicaltrials.gov">http://www.Clinicaltrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

## **Certificate of Confidentiality**

To help us protect your privacy, we have obtained a Certificate of Confidentiality. The researchers can use this Certificate to legally refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

You should also know that there are several circumstances in which the Certificate does not provide coverage. These include when information:

- will be used for auditing or program evaluation internally by the NIH; or
- must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA).
- is necessary for your medical treatment and you have consented to this disclosure;
- is for other research.

In addition, identifiable, sensitive information protected by this Certificate cannot be admissible as evidence or used for any purpose in any action, suit, or proceeding without your consent.

You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

The Certificate of Confidentiality will not protect against the required reporting by hospital staff of information on suspected child abuse, reportable communicable diseases, and/or possible threat of harm to self or others.

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

MEDICAL RECORD

CONTINUATION SHEET for either:

NIH 2514-1, Consent to Participate in A Clinical Research Study

NIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study

STUDY NUMBER: 18-C-0057 CONTINUATION:  pages

### **Stopping Therapy**

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if your disease comes back during treatment
- if you need to take any medications that are prohibited in this study
- if your doctor decides to end the study
- if you become pregnant
- if you have side effects from the treatment that your doctor thinks are too severe
- if new information shows that another treatment would be better for you

In this case, you will be informed of the reason therapy is being stopped.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to Selecta Biosciences, Inc. or designated representatives. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases cannot be recalled and destroyed.

#### **Conflict of Interest**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a Protocol Review Guide. You may ask your research team for a copy of the Protocol Review Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines but they do not need to report their personal finances to the NIH.

Members of the research team working on this study may have up to \$15,000 of stock in the companies that make products used in this study. This is allowed under federal rules and is not a conflict of interest.

The National Institutes of Health and the research team for this study have developed a drug being used in this study. This means it is possible that the results of this study could lead to payments to NIH scientists and to the NIH. By law, government scientists are required to receive such payments for their inventions. You will not receive any money from the development of LMB-100.

PATIENT IDENTIFICATION

#### **CONTINUATION SHEET for either:**

NIH-2514-1 (07-09) NIH-2514-2 (10-84) P.A.: 09-25-0099

| MEDICAL RECORD | N | CONTINUATION SHEET for either: IIH 2514-1, Consent to Participate in A Clinical Research Study IIH 2514-2, Minor Patient's Assent to Participate In A Clinical Research Study |
|---|---|---|
| STUDY NUMBER: | 18-C-0057 | CONTINUATION: pages |

The National Institutes of Health and the research team for this study are using a drug developed by Selecta Biosciences, Inc. through a joint study with your researchers and the company. The company also provides financial support for this study.

## Use of Specimens and Data for Future Research

To advance science, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. A researcher who wants to study the information must apply to the database and be approved. Researchers use specimens and data stored in scientific databases to advance science and learn about health and disease.

We plan to keep some of your specimens and data that we collect and use them for future research and share them with other researchers. We will not contact you to ask about each of these future uses. These specimens and data will be stripped of identifiers such as name, address or account number, so that they may be used for future research on any topic and shared broadly for research purposes. Your specimens and data will be used for research purposes only and will not benefit you. It is also possible that the stored specimens and data may never be used. Results of research done on your specimens and data will not be available to you or your doctor. It might help people who have cancer and other diseases in the future.

If you do not want your stored specimens and data used for future research, please contact us in writing and let us know that you do not want us to use your specimens and/or data. Then any specimens that have not already been used or shared will be destroyed and your data will not be used for future research. However, it may not be possible to withdraw or delete materials or data once they have been shared with other researchers.

#### MEDICAL RECORD

#### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

• Adult Patient or

• Parent, for Minor Patient

STUDY NUMBER:

18-C-0057

CONTINUATION:  pages

## OTHER PERTINENT INFORMATION

1. Confidentiality. When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

The Federal Privacy Act protects the confidentiality of your NIH medical records. However, you should know that the Act allows release of some information from your medical record without your permission, for example, if it is required by the Food and Drug Administration (FDA), members of Congress, law enforcement officials, or authorized hospital accreditation organizations.

- 2. Policy Regarding Research-Related Injuries. The Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the National Institutes of Health, the Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.
- **3. Payments.** The amount of payment to research volunteers is guided by the National Institutes of Health policies. In general, patients are not paid for taking part in research studies at the National Institutes of Health. Reimbursement of travel and subsistence will be offered consistent with NIH guidelines.
- **4. Problems or Questions.** If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Raffit Hassan, M.D., Building 10, Room 4-5330, Telephone: 240-760-6232. You may also call the Clinical Center Patient Representative at 301-496-2626. If you have any questions about the use of your specimens or data for future research studies, you may also contact the Office of the Clinical Director, Telephone: 240-760-6070.
- **5.** Consent Document. Please keep a copy of this document in case you want to read it again.

PATIENT IDENTIFICATION

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)

• Adult Patient or

• Parent, for Minor Patient

NIH-2514-1 (07-09) P.A.: 09-25-0099

MEDICAL RECORD

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

Adult Patient or

• Parent, for Minor Patient

STUDY NUMBER:

18-C-0057

CONTINUATION:  pages

| COMPLETE APPROPRIATE ITEM(S) BELOW: | | | |
|---|---|---|---|
| A. Adult Patient's Consent | | B. Parent's Permission for Minor Patient. | |
| I have read the explanation about this study<br>and have been given the opportunity to discuss<br>it and to ask questions. I hereby consent to<br>take part in this study. | | I have read the explanation about this study<br>and have been given the opportunity to discuss<br>it and to ask questions. I hereby give<br>permission for my child to take part in this<br>study. | |
| | | (Attach NIH 2514-2, Minor's Assorblicable.) | ent, if |
| Signature of Adult Patient/ Legal Representative | Date | Signature of Parent(s)/ Guardian | Date |
| Print Name | | Print Name | |
| C. Child's Verbal Assent (If Appl | icable) | | |
| The information in the above consent was described to my child and my child agrees to participate in the study. | | | |
| Signature of Parent(s)/Guardian | Date | Print Name | |
| THIS CONSENT DOCUMENT HAS BEEN APPROVED FOR USE FROM JANUARY 07, 2019 THROUGH FEBRUARY 04, 2020. | | | |
| Signature of Investigator | Date | Signature of Witness | Date |
| Print Name | | Print Name | |

PATIENT IDENTIFICATION

# **CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)**

• Adult Patient or NIH-2514-1 (07-09)

• Parent, for Minor Patient

P.A.: 09-25-0099